CLINICAL TRIAL: NCT02867956
Title: A Phase II Study of Apatinib In Combination With Etoposide in Patients With Platinum Resistant or Refractory Ovarian Cancer
Brief Title: Apatinib and Etoposide in Patients With Platinum Resistant or Refractory Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xin Huang, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2016-020-01
Record Dates: First submitted 2016-08-03; First posted 2016-08-16 (Estimated); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Ovarian Cancer
Keywords: Ovarian cancer; Apatinib; Etoposide; Chemotherapy
MeSH Terms: conditions — Ovarian Neoplasms | interventions — apatinib; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Apatinib + Etoposide (Experimental): Apatinib 500mg daily, po, and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent.
  Etoposide 50mg daily, po, day 1 to day 14, repeat every 21 days for 6 cycles.
  Interventions: Drug: Apatinib; Drug: Etoposide

INTERVENTIONS:
Drug: Apatinib — Apatinib 500mg daily, po, and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent.
  Other Names: Apatinib mesylate tablets; Aitan
Drug: Etoposide — Etoposide 50mg daily, po, day 1 to day 14, repeat every 21 days for 6 cycles
  Other Names: VP-16

SUMMARY:
The purpose of the study is to evaluate the efficacy and toxicity of apatinib in patients with platinum resistant or refractory ovarian cancer when combined with etoposide.

DETAILED DESCRIPTION:
Ovarian cancer is the leading cause of death for patients with gynecologic malignancies. In most cases, the disease is diagnosed at an advanced stage and approximately 75% of patients will eventually experience disease recurrence. However, the overall response rates of second-line chemotherapy for recurrent ovarian cancer are only 20-27%. Therefore, it is important to seek alternative agent that can improve the outcome. Apatinib is a novel vascular endothelial growth factor receptor 2 tyrosine kinase inhibitor and it has been approved for the treatment of advanced gastric cancer. The preclinical studies suggest apatinib may be effective in other cancers such as ovarian cancer. Therefore, the purpose of this study is to test the efficacy and safety of the study drug apatinib when combined with a standard treatment, etoposide, for patients with platinum resistant or refractory ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or pathologically confirmed diagnosis of epithelial carcinoma of the ovary.
* Platinum resistant ovarian cancer (defined as relapsing within 6 months after the last administration of platinum-based chemotherapy) OR platinum refractory ovarian cancer (defined as progressing while on a platinum-based chemotherapy)
* At least treated with one line of platinum-based chemotherapy
* Female, age ≥18 years and ≤70 years, signed informed consent.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 version
* Patients must have a life expectancy of at least 3 months.
* Patients must have adequate organ function as defined by the following criteria:

  * White blood cell count ≥ 3 x 10^9/L, Absolute neutrophil count (ANC) (≥ 1.5 x 10^9/L), Hemoglobin of ≥ 80 g/L, Platelets ≥ 70 x 10^9/L
  * Total bilirubin ≤ 1 x upper limit of normal (ULN), AST and ALT ≤ 2 x ULN
  * Serum creatinine ≤ 1 x ULN

Exclusion Criteria:

* Had prior exposure to apatinib or has known allegies to any of the excipients.
* History of myocardial infarction, or unstable angina, or New York Heart Association (NYHA) Grade III-IV within 6 months prior to Day 1.
* Patients with QT interval prolongation
* Serious, non-healing wound, active ulcer, bowel obstruction.
* History of abdominal fistula or gastrointestinal perforation within 28 days prior to Day 1
* Evidence of bleeding diathesis or coagulopathy
* Inadequately controlled hypertension
* Major surgical procedure within 28 days prior to Day 1
* Symptomatic central nervous system (CNS) metastasis

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2016-08-10 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2019-09-10 (Actual)

PRIMARY OUTCOMES:
Objective response rate | Up to three years
  Objective response rate defined as confirmed complete response or partial response under RECIST 1.1 criteria. CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. To be assigned a status of CR or PR, changes in tumor measurements must be confirmed by repeat assessments performed no fewer than 4 weeks after the response criteria are first met.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to three years
  Progression-free survival estimated using Kaplan-Meier methods is defined as the time from registration to the earlier of death or disease progression. Patients alive without disease progression are censored at the date of last disease evaluation. Progressive disease (PD) based on RECIST 1.1 is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Equivocal progression of non-target lesions also qualifies as PD.
Duration of Response | Up to three years
  Duration of response was defined as the interval between the date of the first documented response by RECIST 1.1 to the date of first disease progression or death, whichever occurred earlier.
Frequency and severity of adverse effects as defined by CTCAE version 4.03 | 30 days after last dose
  Evaluation of adverse event rate according to CTCAE v4.03
Overall survival (OS) | Up to three years
  Overall survival is defined as the duration from date of enrollment to the date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Huang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Huang X, Xie C, Tang J, He W, Yang F, Tian W, Li J, Yang Q, Shen J, Xia L, Lan C. Adipose tissue area as a predictor for the efficacy of apatinib in platinum-resistant ovarian cancer: an exploratory imaging biomarker analysis of the AEROC trial. BMC Med. 2020 Oct 5;18(1):267. doi: 10.1186/s12916-020-01733-4. PMID 33012286
- [Derived] Lan CY, Wang Y, Xiong Y, Li JD, Shen JX, Li YF, Zheng M, Zhang YN, Feng YL, Liu Q, Huang HQ, Huang X. Apatinib combined with oral etoposide in patients with platinum-resistant or platinum-refractory ovarian cancer (AEROC): a phase 2, single-arm, prospective study. Lancet Oncol. 2018 Sep;19(9):1239-1246. doi: 10.1016/S1470-2045(18)30349-8. Epub 2018 Aug 3. PMID 30082170